CLINICAL TRIAL: NCT06245564
Title: Effect of Ketamine, Amitriptyline and Their Combination on Histaminergic and Non-histaminergic Itch
Brief Title: Effect of Ketamine, Amitriptyline and Their Combination on Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Assistant Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20230046
Record Dates: First submitted 2024-01-25; First posted 2024-02-07 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-10

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — Amitriptyline; Ketamine; Histamine

STUDY DESIGN:
Intervention Model Description: In each participant, the four different creams will be applied in a randomized position. After the cream removal, itch will be induced using histamine in one session and cowhage in the other session.
Masking Description: The participant will be blinded about which cream is applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cream application (Experimental): This subproject will be conducted in two sessions one week apart. Each session will last approximately 3 hours. In each forearm of the participant, two 4x4 cm areas will be selected as Area of Interest (AOI). In these selected areas, the four different creams will be applied in a randomized position for 1½ hours. After the cream removal, itch will be induced using histamine in one session and cowhage in the other session (the order of histamine and cowhage will be randomized). During the application of the substances, the itch/pain elicited will be monitored for 10 minutes using a VAS (Visual analog scale). After the removal of the substances, measurements of SBP, TP, MEI, MPT, MPS, and thermal sensitivity will be conducted.
  Interventions: Drug: Ketamine 0.5%; Drug: Amitriptyline; Drug: ketamine + amitriptyline; Other: Vehicle; Other: Histamine; Other: Cowhage

INTERVENTIONS:
Drug: Ketamine 0.5% — Ketamine cream 0.5% will be applied in a 4x4 area in the forearm of each participant.
Drug: Amitriptyline — Amitriptyline cream 1% will be applied in a 4x4 area in the forearm of each participant.
Drug: ketamine + amitriptyline — A cream containing ketamine 0.5%, amitriptyline 1%, will be applied in a 4x4 area in the forearm of each participant.
Other: Vehicle — A vehicle cream will be applied in a 4x4 area in the forearm of each participant.
Other: Histamine — After the cream removal, itch will be induced using histamine in the first session
Other: Cowhage — After the cream removal, itch will be induced using cowhage in the second session

SUMMARY:
Chronic itch affects approximately a fifth of the global population and is associated with substantial negative consequences for the affected individuals. Furthermore, there is a lack of efficient treat-ment options for chronic itch. Topical ketamine cream has been used successfully to relieve various forms of pain, and we hypothesize that topical ketamine relieves itch through a mechanism of action comparable to that in pain relief.

The aim of this project is to evaluate the effects of ketamine both alone and in combination with amitriptyline on histaminergic and non-histaminergic itch induced by histamine and cowhage, respectively.

DETAILED DESCRIPTION:
The main action of ketamine, 2-(2-chlorophenyl)-2-(methylamino)-cyclohexanone, is to antagonize the glutamate N-methyl-D-aspartate (NMDA) receptors. In the clinical setting, topical ketamine cream has been used successfully to relieve various pathogenic forms of pain. In addition to its pain-relieving effects, the cream was also reported to have itch-relieving properties in a very limited study. However, its efficacy on itch has not been established, and the mechanism of action remains uncertain. Ketamine cream is used not only by itself, but also in conjunction with other analgesics. One of these is amitriptyline, which may enhance the analgesic effects of ketamine. The aim of this human experimental study is to use the well-characterized anesthetic Ketamine, both alone and in combination with amitriptyline, as a tool to modulate different histaminergic and non-histaminergic itch modalities evoked by histamine and cowhage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other drugs
* Previous or current history of neurological, dermatological, immunological, musculoskeletal, cardiac disorder or mental illnesses (psychiatric diagnosis) that may affect the results (e.g., neuropathy, muscular pain in the upper extremities, anxiety, depression, schizophrenia etc.)
* Moles, wounds, scars, or tattoos in the area to be treated or tested
* Current use of medications that may affect the trial such as antihistamines and pain killers.
* Participants had known allergy/discomfort to ketamine or amitriptyline
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain and itch
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical studies)
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Measuring itch by computerized Visual Analog Scale Scoring | Immediately after the intervention
  We will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".
Measuring pain by computerized Visual Analog Scale Scoring | Immediately after the intervention
  We will ask the subjects to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".

SECONDARY OUTCOMES:
Superficial blood perfusion | Immediately after the intervention
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Touch Pleasantness | Immediately after the intervention
  Pleasant touch sensation measured using a standardized sensory brush exerting a force of 200 to 400 mN.
Mechanically evoked itch (MEI), intensity approach | Immediately after the intervention
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Mechanically evoked itch, spatial approach | Immediately after the intervention
  The von-Frey filament that better evokes the itch sensation during the assessment of mechanically evoked itch as well as a template of soft plastic are used to map the area of hyperkinesis in the test areas (forearms).
Mechanical Pain Thresholds (MPT) | Immediately after the intervention
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Sensitivity (MPS), intensity approach | Immediately after the intervention
  This test is conducted with the same pinprick set used to test the MPT.
Mechanical Pain Sensitivity (MPS), spatial approach | Immediately after the intervention
  The pinprick that was selected in the MPT as well as a template of soft plastic are used to map the area of hyperalgesia in the test areas (forearms).
Cold Detection Thresholds (CDT) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thresholds (HPT) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Neuroplasticity and Pain Faculty of Medicine, Aalborg University, Gistrup, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No